CLINICAL TRIAL: NCT02257619
Title: A Randomized, Phase 2 Study of INCB039110 or Placebo in Combination With Docetaxel in Subjects With Previously Treated Stage IIIb, IV, or Recurrent Non-Small Cell Lung Cancer
Brief Title: Study of INCB039110 in Combination With Docetaxel in Subjects With Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to not initiate part 2 due to slow enrollment and competing trials.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 39110-203
Record Dates: First submitted 2014-09-26; First posted 2014-10-06 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: NSCLC (Non-small Cell Lung Carcinoma)
Keywords: Stage IIIb, IV, or Recurrent Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — itacitinib; INCB039110; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Itacitinib plus docetaxel (Experimental)
  Interventions: Drug: Itacitinib; Drug: docetaxel

INTERVENTIONS:
Drug: Itacitinib — Itacitinib tablets administered orally at 400 mg QD for Part 1 of the study.
  Other Names: INCB039110
Drug: docetaxel — Administered as an intravenous infusion in the clinic at 75 mg/m^2 Q3W for Part 1 of the study.

SUMMARY:
The primary objectives of this study is to evaluate the safety and tolerability of itacitinib in combination with docetaxel and to select doses for further evaluation (Part 1, safety run-in portion).

DETAILED DESCRIPTION:
Sponsor decision to not initiate part 2 of the trial and Part 2 of the study was not conducted.

In Part 2, the randomized portion, the objective is to evaluate and compare the overall survival of subjects with previously treated advanced or metastatic non-small cell lung cancer (NSCLC) when treated with itacitinib in combination with docetaxel versus docetaxel alone.

The secondary objectives of this study (Part 2) are to evaluate and compare the efficacy of the 2 treatment groups with respect to progression-free survival, overall tumor response, and duration of response, and to evaluate and compare disease control, safety, and tolerability of itacitinib in combination with docetaxel versus docetaxel alone.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of NSCLC that is Stage IIIb, IV, or recurrent.
2. Received only 1 prior systemic chemotherapy regimen for Stage IIIb, IV, or recurrent disease not including neoadjuvant and/or adjuvant therapy. (NOTE: Exceptions may be allowed based on prior treatment regimens and tumor types in agreement with protocol requirements.)
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
4. Life expectancy of ≥12 weeks.

Exclusion Criteria:

1. Received prior treatment with docetaxel.
2. Known active central nervous system (CNS) metastases. Subjects with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for at least 1 month prior to study entry, defined as:

   1. No evidence of new or enlarging CNS metastasis or new neurological symptoms attributable to CNS metastases.
   2. Subjects who are receiving concomitant corticosteroids must be on a stable or decreasing dose for at least 4 weeks prior to first dose of study treatment and off all anticonvulsants for at least 4 weeks prior to study entry.
3. Peripheral neuropathy ≥ Grade 3.
4. Current or previous other malignancy within 2 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive malignancy.
5. Significant, concurrent, uncontrolled medical condition including but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, cerebral, or psychiatric disease.
6. Unwilling to be transfused with blood components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) | Baseline through 21 days; the end of cycle 1.
  Number of participants with DLT for the determination of the Maximum Tolerated Dose (MTD).

CONTACTS AND LOCATIONS:
Overall Officials: Amit Pande, M.D., Study Director — Incyte Corporation
Locations (16):
- United States (16):
  - Hot Springs, Arizona
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Detroit, Michigan
  - Pascagoula, Mississippi
  - Kansas City, Missouri
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Goldsboro, North Carolina
  - Cleveland, Ohio
  - Gettysburg, Pennsylvania
  - Hershey, Pennsylvania
  - Pawtucket, Rhode Island
  - Spartanburg, South Carolina
  - Round Rock, Texas